CLINICAL TRIAL: NCT05890261
Title: Cooling During Exercise in the Heat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HE2023-0101
Record Dates: First submitted 2023-05-17; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Body Surface Cooling Methods
Keywords: hyperthermia prevention; liquid-perfused cooling garments; mental performance; physical performance

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young healthy subjects (Experimental): Young healthy subjects
  Interventions: Device: Cold water-perfused cooling garment

INTERVENTIONS:
Device: Cold water-perfused cooling garment — Two types of cooling garments will be used. One is a cooling vest and the other includes cooling pants.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of upper-body surface cooling with whole-body surface cooling on exercise performance while wearing firefighter clothing in the heat. The main question it aims to answer is:

• which cooling protocol best prevents an increase in core temperature during exercise in the heat?

Participants will be asked to participate three times in a 60-minute exposure (to 40 degrees C, 40% relative humidity) in which they conduct three work/rest periods including 15 minutes of stepping exercise (20 steps/minute) and 5 minutes of rest. The following three conditions will include:

* Control: no cooling garments
* Upper-body cooling: cold water-perfused cooling vest
* Whole-body cooling: cold water-perfused cooling pants and cooling vest

DETAILED DESCRIPTION:
The objectives are to determine thermoregulatory stress (e.g., change in skin and core temperature), physiologic stress (e.g., heart rate and metabolism), cognitive function (Mini-Cog; includes clock drawing and three-word recall), and subjective responses (e.g., thermal comfort, heat sensation, rating of perceived exertion, subjective wetness, breathing comfort) during three conditions while exercising in the heat while wearing thermal protective clothing. The conditions are control (no cooling), upper-body cooling, and whole-body cooling.

Physiologic measures:

Core temperature. Core temperature (°C) will be monitored with e-Celsius, an ingestible pill that continuously monitors, records, and wirelessly transmits core temperature.

Skin temperature. Mean skin temperature (ºC) will be measured with small metal discs (iButton, EDS) taped to the skin at the following 7 sites: forehead, chest, abdomen, upper arm, lower arm, anterior thigh, and anterior calf.

Heart rate and respiration. A Hexoskin shirt will be worn. Sensors in the shirt measure heart rate and chest expansion for breathing indicators.

Metabolism. Subjects will wear a face mask and oxygen consumption, VCO2 and minute ventilation is going to be continuously monitored with a metabolic cart.

Sweat loss. Will be determined from differences in body and clothing weight measured before and after the exercise trials.

Subjective measures:

Every 20 minutes during the exercise test (see below), participants will be asked to rate the following: thermal comfort, heat sensation, rating of perceived exertion (RPE), breathing comfort, and skin wetness.

This will be followed by a test of cognitive function. This involves two components: a three-item recall test and a clock-drawing task. Investigators will ask the subject to repeat three unrelated words (e.g., apple, table, penny) and then will ask them to recall those words after a few minutes. While the subject is trying to recall the words, investigators will ask them to draw a clock face including all of the numbers, and the hands showing a specific time (e.g., 10 minutes past 11). Then the subjects will then be asked to repeat the original 3 words in order.

Cooling procedures:

Cooling will be applied through a liquid-perfused shirt and pants. Each garment has small tubes sewn into the interior of the garment. Cold water (3-8 degrees C) will be perfused through the garments at 5 l/min. The garments will be worn over the Hexoskin shirt and shorts.

Exercise test:

This 60-minute test involves 3 sets of 15 minutes of stepping exercises (20 steps per minute) followed by 5 minutes of sitting rest. During the rest periods, They will be asked to give their subjective evaluations of thermal comfort, heat sensation, rating of perceived exertion, breathing comfort, skin wetness, and cognitive function.

The exercise test will be stopped and the subject will exit the chamber if: the core temperature reaches 39 degrees C; the subject feels light-headed, or nausea; the subject indicates a wish to stop for any reason; or a researcher feels the subject should stop for any reason.

Protocol:

Once subjects have been instrumented they will sit for 10 minutes of baseline measurements in the laboratory (~20 degrees C). They will then enter a climatic chamber (40 degrees C, 40% humidity) and complete the 60-minute exercise/rest protocol. They will then exit the chamber and sit for another 10 minutes of post-exercise measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years.
* Meet the criteria on the CSEP Get Active Questionnaire
* Answer 'no' to questions in the Screening Questionnaire.

Exclusion Criteria:

* Outside the accepted age bracket.
* Not meeting the criteria on the CSEP Get Active Questionnaire or the Screening Questionnaire.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Core temperature | Times 0, 30, 50, 70 and 85 min
  Core temperature will be measured with a radio pill that is ingested 2 hours pre-trial.

SECONDARY OUTCOMES:
Change in Mental performance | Times 0, 30, 50, 70 and 85 min
  Mini-Cog test for recall and cognition

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (1):
- 211 Max Bell Centre, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No